CLINICAL TRIAL: NCT00032149
Title: Pilot Study Of PMitCEBO Plus G-CSF In Good-Prognosis HIV-Related Lymphoma
Brief Title: Combination Chemotherapy Plus Filgrastim in Treating Patients With HIV-Related Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lymphoma Trials Office (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000069261; BNLI-GOODRISKHIV; EU-20144
Record Dates: First submitted 2002-03-08; First posted 2003-01-27 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2007-03

CONDITIONS: Lymphoma
Keywords: AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; AIDS-related diffuse large cell lymphoma; AIDS-related immunoblastic large cell lymphoma; AIDS-related small noncleaved cell lymphoma; AIDS-related diffuse mixed cell lymphoma; AIDS-related diffuse small cleaved cell lymphoma; AIDS-related lymphoblastic lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Bleomycin; Filgrastim; Cyclophosphamide; Etoposide; Mitoxantrone; Prednisolone; Vincristine

INTERVENTIONS:
Biological: bleomycin sulfate
Biological: filgrastim
Drug: cyclophosphamide
Drug: etoposide
Drug: mitoxantrone hydrochloride
Drug: prednisolone
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells. Colony-stimulating factors such as filgrastim may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of chemotherapy.

PURPOSE: Phase I/II trial to study the effectiveness of combining filgrastim with combination chemotherapy in treating patients who have HIV-related non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicity of mitoxantrone, cyclophosphamide, etoposide, vincristine, bleomycin, prednisolone, and filgrastim (G-CSF) in patients with good-prognosis (defined by the study as having 1 adverse prognostic factor) HIV-related non-Hodgkin's lymphoma.
* Determine the effects of this regimen on response rate, time to disease progression, and survival in these patients.

OUTLINE: This is a multicenter study.

Patients receive mitoxantrone IV, cyclophosphamide IV, and etoposide IV on day 1; and vincristine IV and bleomycin IV on day 8. Patients also receive prednisolone daily on weeks 1-4 and then every other day on weeks 5-16. Patients receive filgrastim (G-CSF) subcutaneously on days 6-12. Treatment repeats every 2 weeks for up to 8 courses (16 weeks) in the absence of disease progression or unacceptable toxicity. Patients with complete response (CR) or partial response (PR) receive 4 courses beyond CR or PR.

Patients are followed every 3 months for 1 year, every 6 months for 5 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 15-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed previously untreated HIV-related non-Hodgkin's lymphoma with 1 of the following:

  * Prior diagnosis of acquired immune deficiency syndrome (AIDS)
  * CD4 count < 100,000/mm3
  * ECOG performance status > 2

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* See Disease Characteristics

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Not specified

Renal:

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic:

* Not specified

Chemotherapy:

* Not specified

Endocrine:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2001-10

PRIMARY OUTCOMES:
Toxicity
Effects of treatment on response rate, time to disease progression, and survival

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Pettengell, MD, Study Chair — St George's, University of London
Locations (4):
- United Kingdom (4):
  - Cheltenham General Hospital, Cheltenham, England
  - St. Georges, University of London, London, England
  - King's College Hospital, London, England
  - Edinburgh Cancer Centre at Western General Hospital, Edinburgh, Scotland